CLINICAL TRIAL: NCT06361186
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Phase I Study to Evaluate the Tolerability, Pharmacokinetics and Pharmacodynamics of Proximod in Healthy Subjects.
Brief Title: Proximod Pharmacokinetics In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longevity Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJXH-2017-001
Record Dates: First submitted 2024-03-12; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet, qd, oral administration for 28 days
  Interventions: Drug: Placebo
- test drug (Experimental): Proximod Tablets, 6mg and 12mg, qd, oral administration for 28 days
  Interventions: Drug: Proximod

INTERVENTIONS:
Drug: Proximod — Single and multiple-dose to establish the safety and PK profile
  Other Names: IMM-H001
  Arms: test drug
Drug: Placebo — Placebo controlled
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the tolerability, pharmacokinetics and pharmacodynamics of Proximod in healthy subjects. The main questions it arms to answer are:

1. to evaluate the safety and tolerance of Proximod in healthy subjects after single or repeated doses.
2. to learn the pharmacodynamics of Proximod in healthy subjects after single or repeated doses.
3. to evaluation of the effect of food on the pharmacokinetics of Proximod in healthy subjects Participants will receive test tablets or placebo at the indicated date and collect blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Before the test, sign an informed consent form and fully understand the written test content, process and possible adverse reactions.
* Complete research in accordance with the requirements of the trial plan.
* Subjects (including partners) are willing to have no pregnancy plans in the next 6 months and voluntarily take effective contraceptive measures.
* Male and female subjects aged 18 to 50 years old (including 18 and 50 years old).
* Male subjects must weigh no less than 50 kg, and female subjects must weigh no less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), body mass index is in the range of 18~28kg/m2 (including the critical value).
* Health status: No clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system (such as asthma, exercise-induced asthma, chronic obstructive pulmonary disease), mental disorder, metabolic abnormality, etc.
* Normal physical examination and vital signs or abnormal without clinical significance.

Exclusion Criteria:

* Those who smoked more than 5 cigarettes per day in the 3 months before the test.
* Have a history of allergy to the trial drug or its excipients, or allergic constitution (allergy to multiple drugs and food).
* Have a history of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine).
* Blood donation or significant blood loss (>450 mL) within three months before screening.
* Taking any drugs that alter liver enzyme activity 28 days before screening.
* Take any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines within 14 days before screening.
* Those who have taken special diets (including dragon fruit, mango, grapefruit, etc.) or engaged in strenuous exercise within 2 weeks before screening, or other factors that affect drug absorption, distribution, metabolism, excretion, etc.
* Concomitant inhibitors or inducers of CYP3A4, P-gp or Bcrp such as itraconazole, ketoconazole or dronedarone.
* Recent significant changes in eating or exercise habits.
* Participated in a drug clinical trial within three months before taking the study drug.
* Have a history of dysphagia or any gastrointestinal disease that affects drug absorption.
* Suffering from any disease that increases the risk of bleeding, such as acute gastritis or gastric and duodenal ulcers.
* ECG abnormalities have clinical significance or QTC>470ms in men or QTC>480ms in women.
* Abnormal and clinically significant ophthalmic examination, including fundus examination, optical coherence tomography.
* Female subjects are lactating or have positive serum pregnancy results during the screening period or during the trial.
* Clinically significant abnormalities in clinical laboratory tests or other clinically significant following diseases diagnosed within 12 months (including but not limited to gastrointestinal, renal, liver, neurological, blood, endocrine, tumor, lung, immune, psychiatric or Cardiovascular disease).
* Positive screening results for viral hepatitis (including hepatitis B and hepatitis C), HIV antibodies, and Treponema pallidum antibodies.
* Acute illness or concomitant medication occurs from the screening stage to study medication.
* Ingested chocolate, any caffeinated or xanthine-rich food or drink 24 hours before taking study drug.
* Positive alcohol breath test 24 hours before taking study medication or upon check-in.
* Those with a positive urine drug screen or a history of drug abuse within the past five years or 3 years before the test.
* Intolerance to standard meals (two boiled eggs, a piece of toast with buttered bacon, a box of fried potato chips, a glass of whole milk).
* Subjects (this article only applies to subjects participating in postprandial trials).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 64 days
Time to peak plasma concentration (Tmax) | Up to 64 days
The lowest plasma concentration (Cmin) | Up to 64 days
Half-life (t1/2) | Up to 64 days
Number of adverse events and number of participants with adverse events | Up to 64 days

SECONDARY OUTCOMES:
Lymphocyte count | Up to 64 days
Percentage of CD3+CD4+ and CD3+CD8+ T cells | Up to 64 days

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Li Q, Li C, Wu M, Chen H, Li Y, You F, Zhao Y, Jin J, Chen X, Ding Y. Evaluation of proximod, a selective agonist of sphingosine-1-phosphate receptor-1, in healthy volunteers and patients with rheumatoid arthritis: a phase 1, double-blind, randomised, placebo-controlled, ascending dose trial. Lancet Rheumatol. 2024 Dec;6(12):e837-e847. doi: 10.1016/S2665-9913(24)00199-1. Epub 2024 Oct 22. PMID 39454617